CLINICAL TRIAL: NCT02503618
Title: Understanding Substance Use and Incident HIV/STI Among Young Black Men Having Sex With Men (MSM)
Brief Title: Understanding Substance Use and Incident HIV/STI Among Young Black MSM
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Other Study IDs: IRB00078950; 1R01DA038196-01 (NIH)
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: HIV; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spot testing, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-negative YBMSM: Subjects are young black men who have sex with men in Atlanta, Georgia and are HIV-negative
- HIV-positive YBMSM: Subjects are young black men who have sex with men in Atlanta, Georgia and are HIV-positive

SUMMARY:
The scientific purpose of this study is to look at how substance use may relate to human immunodeficiency virus (HIV) infection among young black men who have sex with men in Atlanta.

DETAILED DESCRIPTION:
Young black men who have sex with men (YBMSM) are a critically at-risk population in the United States and Atlanta that faces extremely high incidence rates of HIV and other sexually transmitted infections (STIs). The understanding of what places this group of men at high risk is incomplete, and the role of substances in amplifying that risk is unclear. This study will fill a number of gaps about how substances and partnerships place YBMSM at increased HIV risk. The study includes several innovative aspects. First, the investigators are using a theoretical framework to understand multilevel associations between substance use and HIV risk behavior in YBMSM in the southeastern United States, a critically at-risk but understudied population. Second, the investigators are using a variety of enhanced measurement methods to understand these associations. The investigators are supplementing self-reported substance use with objective measures to enhance the sensitivity of classifying recent use. The investigators will analyze incident HIV/STI endpoints in addition to self-reported sexual behaviors. The investigators will use detailed, event-based and dyadic measures of substance use and its covariates, which will capture both sexual and non-sexual contexts of use. Although previous cohort studies have explored alcohol and drug use during sexual events among men who have sex with men (MSM), few studies have described both sexual and non-sexual patterns of, and motivations for, substance use among YBMSM, and none have incorporated longitudinal biomarkers of substance use and related these to incident infection outcomes. Finally, the investigators are using a mixed-methods approach to provide context to the quantitative findings. By recruiting subjects to a nested qualitative study within the larger cohort based on their interval-specific risks, the investigators will gain in-depth information regarding the emergence, persistence, and resolution of these complex relationships between substances and sexual risk behaviors among YBMSM and how these relationships emerge and are resolved over time.

ELIGIBILITY:
Inclusion Criteria:

* male at birth
* currently identifies as male
* age ≥18 years and < 30 years at enrollment
* had anal sex with a man in lifetime
* has had any sex with a man in the past 3 months
* self-reported race is black/African American
* lives in Atlanta area and plans to remain for 2 years
* is able to complete the survey instruments in English
* is willing to provide at least 2 means of contact
* is willing to be re-contacted for the return of HIV/STI testing results, and for other study reasons as necessary
* is not enrolled in an HIV prevention trial

Exclusion Criteria:

* self-reported multiple or non-Black/African American race(s)
* self-reported Hispanic ethnicity
* (for prospective follow-up) participant screens HIV-positive

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young black men who have sex with men in Atlanta, Georgia will be recruited in a variety of venues in Atlanta. If needed, there will be targeted recruitment via Facebook.
Sampling Method: Non-Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2015-07; Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Hazard ratio for HIV incidence and levels of alcohol, marijuana, cocaine, and ecstasy use | 2 years
  Prevalence of drug use and association between these factors and HIV seroconversion (hazard ratio)
Incidence rates of biomarker-detected and self-reported alcohol, marijuana, cocaine, and ecstasy use | 2 years
Proportion of recent sex partners who are additionally substance-use partners | 2.5 years
Incidence rates of HIV | 2 years
  Total person-years will be calculated as the time from study entry to the estimated date of seroconversion.

SECONDARY OUTCOMES:
Event-level odds ratios between serodiscordant unprotected anal intercourse and self-reported alcohol, marijuana, cocaine, and ecstasy use | 2.5 years
Incidence rates of sexually transmitted infections (rectal gonorrhea, rectal chlamydia, urethral gonorrhea, urethral chlamydia, syphilis) | 2 years
  Total person-years will be calculated as the time from study entry to the estimated date of seroconversion.
Rate ratios between sexually transmitted infection (STI) incidence and levels of biomarker-detected and self-reported alcohol, marijuana, cocaine, and ecstasy use | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Sullivan, DVM, PhD, Principal Investigator — Emory University
Locations (7):
- United States (7):
  - Grady Health System, Atlanta, Georgia
  - Grady Infectious Diseases Clinic (Ponce Clinic), Atlanta, Georgia
  - The Ponce de Leon Center of the Grady Health System, Atlanta, Georgia
  - AID Atlanta, Atlanta, Georgia
  - Southside Medical Center, Atlanta, Georgia
  - Rollins School of Public Health, Atlanta, Georgia
  - SisterLove, Inc, Atlanta, Georgia

REFERENCES:
- [Derived] Serota DP, Rosenberg ES, Thorne AL, Sullivan PS, Kelley CF. Lack of health insurance is associated with delays in PrEP initiation among young black men who have sex with men in Atlanta, US: a longitudinal cohort study. J Int AIDS Soc. 2019 Oct;22(10):e25399. doi: 10.1002/jia2.25399. PMID 31592575
- [Derived] Serota DP, Rosenberg ES, Sullivan PS, Thorne AL, Rolle CM, Del Rio C, Cutro S, Luisi N, Siegler AJ, Sanchez TH, Kelley CF. Pre-exposure Prophylaxis Uptake and Discontinuation Among Young Black Men Who Have Sex With Men in Atlanta, Georgia: A Prospective Cohort Study. Clin Infect Dis. 2020 Jul 27;71(3):574-582. doi: 10.1093/cid/ciz894. PMID 31499518
- [Derived] Serota DP, Rosenberg ES, Lockard AM, Rolle CM, Luisi N, Cutro S, Del Rio C, Siegler AJ, Sanchez TH, Sullivan PS, Kelley CF. Beyond the Biomedical: Preexposure Prophylaxis Failures in a Cohort of Young Black Men Who Have Sex With Men in Atlanta, Georgia. Clin Infect Dis. 2018 Aug 31;67(6):965-970. doi: 10.1093/cid/ciy297. PMID 29635415